CLINICAL TRIAL: NCT06885164
Title: Seismocardiographic Monitoring in Heart Failure
Brief Title: Remote Monitoring of Cardiac Mechanics in Heart Failure Patients
Acronym: SeismicHeart
Status: Recruiting | Type: Observational
Sponsor: Aalborg University (Other)
Collaborators: Aalborg University Hospital (Other); Copenhagen University Hospital at Herlev (Other)
Responsible Party: Principal Investigator, Samuel Schmidt, Associate Professor, Aalborg University
Other Study IDs: N-20240038
Record Dates: First submitted 2024-09-10; First posted 2025-03-20 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; Heart Failure - NYHA II - IV
Keywords: heart failure; remote monitoring; cardiac mechanics
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Heart Failure Participants: The included participants will be heart failure patients that are hospitalized or visits a heart failure clinic. The participants should be in NYHA Class II or higher and 18-90 years old. The participant should wear the sensor for 30 days, and it will measure every hour for the 30 days. Moreover, the participant should undergo echocardiography and answer questionnaire at enrollment day and at the last day of the study (day 30).
  Interventions: Other: Continuous monitroing

INTERVENTIONS:
Other: Continuous monitroing — Continuous monitoring for 30 days with a small combined SCG and 1-lead ECG sensor

SUMMARY:
Heart failure is a severe heart disease, where the heart's ability to pump blood is unsatisfactory. The consequence is a high risk of hospitalization and death. Heart failure is treated with medicine which relieves symptoms and slows down the disease progression. This medical treatment needs routine adjustment, but in many cases, this adjustment is not done timely, which results in life treating conditions where the patients need acute hospitalization. Remote health monitoring of HF patients has the potential to ensure timely adjustment. However, only sensors placed inside the blood vessels of the lung, have been shown effective. The disadvantage is that the placement of the sensor requires surgery. This makes the method costly and poses a risk for the patient. The aim of the current project is to develop a small intelligent patch, which can measure the heart's function from the outside of the body. The method will be low-cost, simple to use and will not pose a risk to the patient.

DETAILED DESCRIPTION:
The goal of this observational study is to gather data from heart failure participants, and to investigate whether it is possible to detect early alterations in heart failure based on this data. The main goals are

* Investigate whether parameters extracted from the measured data provide information regarding heart failure alterations
* Investigate if it is possible to detect alterations at early stages

The gathered data will be measured from a little sensor placed on sternum measuring acceleration (seismocardiography (SCG)) and electrocardiography (ECG) to provide an impression of the heart's mechanical function and electrical function, respectively. This data from the sensor will be analyzed with respect to other parameters obtained from, among others, echocardiography, total blood volume, changes in medical therapy, and hospitalization.

The included heart failure participants should be in the age group 18-90 years and in New York Heart Association Functional Classification (NYHA) class II or higher. Participants will wear the sensor to measure the participant's cardiac mechanics and electronics simultaneously. The participants will:

* wear the sensor for a period of 30 days from discharge or visit to heart failure clinic. The sensor will measure SCG and ECG for a short period (less than 30 seconds) once every hour,
* fill out questionnaires at first and last day of the study
* undergo echocardiography at first day and last day of the study
* not change everyday life because of the sensor

ELIGIBILITY:
Inclusion Criteria:

* NYHA Class II or higher
* 18-90 years old

Exclusion Criteria:

* Pregnancy
* Drug addiction defined as the use of cannabis, opioids, or other drugs
* Mechanical heart valves
* In dialysis
* Not possible to obtain clinical echocardiography of sufficient quality
* Lack of ability to coorperate

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be obtained from Aalborg University Hospital or Herlev-Gentofte Hospital in Denmark that are hospitalized or visits the heart failure clinic due to their heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Heart Failure Related Hospitalization | Within 60 days of enrollment
  It will during the study be noted if an enrolled participant is hospitalized due to an alteration in heart failure condition.

SECONDARY OUTCOMES:
Rate and direction of Adjustement in Medical Therapy | During the 30 days
  Adjustments in the use of loop diuretics (furosemide, metolazon, bumetanide and torasemide) will be noted during the study.
Differences in Echocardiographic extracted strain pre and post study period | Day 1 and day 30
  Strain (%) extracted from echocardiography at day 1 and day 30 at the study.
Score of Patient Experience | At day 30
  The participant's experiences using the sensor and compliance using the sensor. This will be obtained through a questionnaire fulfilled by enrolled participants. It is a System Usabaility Scale for use of the sensor. The score will be between 0 and 5. A higher score means better user experience with the system.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Aalborg University Hospital, Aalborg, Denmark
  - Copenhagen University Hospital Herlev, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No